CLINICAL TRIAL: NCT05690139
Title: Evaluation of Bariatric Surgery Patients Before and After Sleeve Gastrectomy in Terms of Protein-energy and Food Groups Consumption by Three Factors Eating Scale and Healthy Eating Index
Brief Title: Evaluation of Bariatric Surgery Patients Before and After Sleeve Gastrectomy in Terms of Nutritional Status
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Other Study IDs: ETK00-2020-0168
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Bariatric Surgery Candidate; Healthy Eating Index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients: Obese patients received LSG surgery approval
  Interventions: Procedure: Pre-operative LSG patients; Procedure: Post-operative patients 1st month; Procedure: Post-operative patients 3rd month; Procedure: Post-operative patients 6th month

INTERVENTIONS:
Procedure: Pre-operative LSG patients — Baseline
Procedure: Post-operative patients 1st month — 1 month after surgery
Procedure: Post-operative patients 3rd month — 3 months after surgery
Procedure: Post-operative patients 6th month — 6 months after surgery

SUMMARY:
Background/purpose: Laparoscopic sleeve gastrectomy (LSG) has been defined as an innovative surgical method for the treatment of obesity and is progressively applied worldwide. However, data on result of sleeve gastrectomy regarding energy-protein status, nutrient deficiencies and body composition are limited. The purpose of this study is to search nutritional status, body composition and biochemical parameters following LSG.

Methods: Obese subjects (N:55) scheduled for sleeve gastrectomy were included. Macro-micronutrient intake analysis, biochemical blood parameters, and anthropometric measures were performed before and 1, 3 and 6 months after LSG.

DETAILED DESCRIPTION:
Background/purpose: Laparoscopic sleeve gastrectomy (LSG) has been defined as an innovative surgical method for the treatment of obesity and is progressively applied worldwide. Nutritional deficiencies are identified as the possible complications of bariatric surgery. However, data on result of sleeve gastrectomy regarding energy-protein status, nutrient deficiencies and body composition are limited. The purpose of this study is to search nutritional status, body composition and biochemical parameters following LSG.

Methods: Obese subjects (N:55) scheduled for sleeve gastrectomy were included in this study. Preoperative and postoperative (1, 3 and 6th months) protein-energy and other nutrient consumptions, eating habits, food consumption diversity were evaluated with food frequency questionnaire, 3-days food diary record, three-factor eating scale and healthy eating index. Also in the pre- and postoperative period; anthropometric (weight, height, waist, hip, fat free mass) values measured and biochemical blood parameters were collected.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* To have sleeve gastrectomy surgery,
* To be over 18 and under 65 years old
* Not having a perception disorder and communication problems

Exclusion Criteria:

* Ages <18 or >65 years old
* Having a pacemaker (implantation) or any prosthesis (inconvenient for segmental body analysis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of patients who received LSG surgery approval which was conducted in a special obesity clinic, Obezite Cerrahi Ankara Merkezi in Ankara, Turkey.
  The decision for surgery was taken after a multidisciplinary meeting, following recommendations of international consensus conferences or expert panels American Society for Metabolic and Bariatric Surgery (ASMBS).
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Comparing the 3-day food diaries (1 weekend day and 2 weekdays) taken during each intervention (pre-post operative 1,3,6 months) | 6 months
  Daily nutrient intake was calculated by using computer software (Stuttgart, Germany; Turkish version: BeBiS, Vers. 9)
Three Factor Eating Questionnaire Revised-21 (TFEQ-Tr21) scale | 6 months
  Dietary Behavior: A modification of the Three Factor Eating Questionnaire (TFEQ-TR21) was used to assess cognitive restraint of eating, disinhibition, and hunger.
Healthy Eating Index (HEI-2010) | 6 months
  Diet Quality: was assessed using the HEI-2010, a measure of diet quality that assesses how well dietary intake aligns with key recommendations.

SECONDARY OUTCOMES:
Comparing the waist circumference (cm) of all interventions | 6 months
  after the pre and post operative intervention waist circumferences (midway between the rib cage and the iliac crest) were measured using a flexible tape.
Comparing the body mass index (BMI) of all interventions | 6 months
  BMI was calculated (weight/height squared; in kilograms per square meter)
Comparing the body fat percentage (%) of all interventions | 6 months
  the percentage of body fat and fat free mass (FFM) was measured by Tanita Segmental Body Composition Analyzer MC-780MA-N.
Comparing the fasting blood glucose levels of all interventions | 6 months
  Concentration of fasting blood glucose levels baseline and changes after 1,3 and 6 months after surgery were compared. Blood samples were obtained from medical files before surgery and after 1,3,6 months of surgery period, and sera were stored at -30∘ C, until analytical measurements were performed.
Comparing the serum lipid levels of all interventions | 6 months
  Differences in concentration of serum lipid levels of participants in baseline period and after post-operation were measured.
  Blood samples were obtained from medical files at baseline period (pre-operation) and after each intervention period (post-operation 1.3.6 months), and sera were stored at -30∘ C, until analytical measurements were performed. The levels of serum lipids: Triglycerides (mg/dL), Total cholesterol (mg/dL), and HDL cholesterol (mg/dL) were determined using a Dimension Xpand Plus integrated clinical chemistry autoanalyzer (Siemens Healthcare Diagnostics, USA).
Comparing the serum B12 levels of all interventions | 6 months
  baseline, 1,3,6, months after surgery B12 blood measurements taken from patients medical files.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Erge, Asst. Prof., Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided